CLINICAL TRIAL: NCT04426084
Title: Cardiovascular Disease, Cardiovascular Risk Factors, Treatments and Severe COVID-19 Outcomes. A Nationwide Registry-based Case-Control Study
Brief Title: Cardiovascular Risk Factors and Severe COVID-19. A Nationwide Registry-based Case-Control Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Per Svensson, Associate professor, Karolinska Institutet
Other Study IDs: 4
Record Dates: First submitted 2020-06-09; First posted 2020-06-11 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Adiposity; Antihypertensive Agents; Hydroxymethylglutaryl-CoA Reductase Inhibitors; Cardiovascular Agents

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Hypertension — Exposure : Any registered diagnosis of I10 within 15 years or a registered pick-up of a prescription of antihypertensive treatment (ATC C02CA, C02DB02, C03, C07, C08, C09) within one year before index date in the Swedish prescribed drug register (exluding those with a registered diagnosis of other indications for betablocker (heart failure, atrial fibrillation) or ACE-inhibitor, ARB(heart failure) ) Exposures will be compared between cases and controls and between cases with different outcomes and controls
Other: Diabetes type 2 — Exposure: Any registered diagnosis of E11 within 15 years or a registered pick-up of a prescription with any antidiabetic treatment (ATC A10) within one year before index date in the Swedish prescribed drug register.
  Exposures will be compared between cases and controls and between cases with different outcomes and controls
Other: Obesity — Exposure: Diagnosis ICD E66 within 15 years before index date Exposures will be compared between cases and controls and between cases with different outcomes and controls
Drug: Antihypertensive Agents — Pick up of a prescription of C02CA, C02DB02, C03, C07, C08, C09 registered in the Swedish prescribed drug register within 6 month before index date.
  Exposures will be studied separately for each antihypertensive class and compared between cases and controls and between cases with different outcomes and controls
Drug: Statins (Cardiovascular Agents) — Pick up of a prescription of C10AA registered in the Swedish prescribed drug register within 6 month before index date.
Other: Chronic kidney disease — Exposure: Diagnosis ICD N18 within 15 years before index date Exposures will be compared between cases and controls and between cases with different outcomes (mechanical ventilation, continuous renal replacement therapy mortality) and controls. Exposures will thereafter be compared in subgroups by BMI at ICU-admission and in subgroups matched by history of type 2 diabetes.

SUMMARY:
In this study we cross-reference several nationwide high-quality Swedish registers in order to study risk factors for severe Covid-19 outcomes.

DETAILED DESCRIPTION:
In this nationwide, case-control study we cross-reference several detailed, high-quality Swedish registers in order to study risk factors associated with severe Covid-19 as well as different disease outcomes, with a focus on cardiovascular disease, chronic kidney disease, different treatments and socioeconomic factors. Cases are identified through the Swedish intensive care register (SIR) and controls through the Swedish population register (RTB). Further information on the study participants is gathered by linkage to registers on: prescribed drugs; history of in- and outpatient care; income, education and migration. Follow-up data such as future hospitalization and mortality will be gathered prospectively.

ELIGIBILITY:
Inclusion Criteria:

* Cases: Admitted to intensive care unit in Sweden and registered admission in the Swedish intensive care register (SIR) with a main diagnosis of Covid-19 confirmed by laboratory testing (ICD10: U07.1). (cases)
* Control subjects matched for age, gender,residency: For each case 10 controls matched for age, gender and district of residence will be identified by Statistics Sweden (SCB) in the Swedish population register (RTB).
* Control subjects matched for age and gender: For each case 5 controls matched for age and gender will be identified by by Statistics Sweden (SCB) in the Swedish population register (RTB).

Exclusion Criteria:

* No valid Swedish personal identity number (PIN)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 1,424 cases and 14,240 control subjects (first analysis june 2020) A total of 4684 cases and 46840 control subjects (july 2022)
Sampling Method: Non-Probability Sample
Enrollment: 22784 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-06-08 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Severe Covid-19 | 2020-03-01 to 2020-05-11
  Admitted to ICU in Sweden with a main diagnosis of Covid-19 confirmed by laboratory testing (ICD 10: U07.1) and requring mechanical ventilation
Severe Covid-19 with pulmonary embolism | 2020-03-01 to 2020-05-11
  Admitted to ICU in Sweden with a diagnosis of Covid-19 confirmed by laboratory testing (ICD 10: U07.1) and a bidiagnosis of pulmonary embolism (ICD10:I26)

SECONDARY OUTCOMES:
CRRT(Continuous Renal Replacement Therapy) | 2020-03-01 to 2020-05-11
  Number of participants admitted to ICU in Sweden with a verified diagnosis of Covid-19 requring CRRT
ECMO (Extracorporeal Membrane Oxygenation ) | 2020-03-01 to 2020-05-11
  Number of participants admitted to ICU in Sweden with a verified diagnosis of Covid-19 requring ECMO
ICU Mortality | 2020-03-01 to 2020-05-11
  Number of participants admitted to ICU in Sweden with a verified diagnosis of Covid-19 with death occurring in ICU after admission

CONTACTS AND LOCATIONS:
Locations (1):
- Södersjukhuset, Stockholm, Sweden

REFERENCES:
- [Derived] Svensson P, Hofmann R, Habel H, Jernberg T, Nordberg P. Association between cardiometabolic disease and severe COVID-19: a nationwide case-control study of patients requiring invasive mechanical ventilation. BMJ Open. 2021 Feb 17;11(2):e044486. doi: 10.1136/bmjopen-2020-044486. PMID 33597145